CLINICAL TRIAL: NCT06992388
Title: The Influence of Shoulder Manipulation on Muscle Strength and Stiffness and Motor Functionality of Volleyball Players During Training
Brief Title: Application Shoulder Manipulation in Volleyball Players
Acronym: Manual Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KB/94/2025
Record Dates: First submitted 2025-05-17; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Manual Therapy; Manipulation; Muscles
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual Therapy; Other: Placebo; Other: Tape elastic
- Group B (Placebo Comparator): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual Therapy; Other: Placebo; Other: Tape elastic
- Group C (Active Comparator): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual Therapy; Other: Placebo; Other: Tape elastic

INTERVENTIONS:
Other: Manual Therapy — This technique involves a low-amplitude, high-velocity push on the shoulder joints with an additional two-second tension
Other: Placebo — This technique involves a low-amplitude, high-velocity push on the shoulder joints with an additional two-second tension
Other: Tape elastic — The following intervention will be performed: application with an elastic band

SUMMARY:
Currently, it is difficult to find studies in the literature assessing the influence of manual therapy on kinetic and kinematic factors for the upper limbs of volleyball players, which in the long run may translate into a reduction in injuries by improving strength and balance in athletes, when planning training or therapy.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals who are over 18 years old,
* a player from the AZS volleyball league,
* a player who regularly competes in the league,
* expressing informed consent to participate in the study and undertaking to comply with the track regulations and wear a helmet.

Exclusion Criteria:

* lack of volunteer consent,
* previous surgeries of the upper, lower limb and spine,
* other upper limb injuries in the last 6 months,
* pain limiting participation in the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of MVC. | The study will be conducted 3 times: pre-intervention, immediately after the intervention and immediately after training session. Each isometric muscle test lasts 3 seconds.
  Muscle EMG is an assessment of electrical characteristics during the test, the electrical source of which is the muscle membrane potential, and measured in μV.
Assessment of MVC. | The study will be conducted 3 times: pre-intervention, immediately after the intervention and immediately after training session.Each isometric muscle test lasts 3 seconds.
  Muscle EMG is an assessment of electrical characteristics during the test, which is measured by the repetition frequency of muscle motor unit discharges, which is measured in Hz, at the same time of the test.Time
Muscle stiffness | The study will be conducted 3 times: pre-intervention, immediately after the intervention and immediately after training session. Each Myoton application lasts 1 sec for one point.
  Muscle stiffness - characteristic resistance to physical contraction, which deforms initially forming. Stiffness (N/m) was calculated as S = amax.mprobe/Δl.

SECONDARY OUTCOMES:
Assessment of proprioception. | The test will be performed 3 times: pre-intervention, immediately after the intervention and immediately after training session. Each joint measurement will be performed at three settings: 30, 45 and 90 degrees.
  Assessing proprioception is an assessment of the angular position of a joint and then an attempt to reproduce it, measured in degrees.
Y balance test | The test will be conducted 3 times: pre-intervention, immediately after the intervention and immediately after training session.
  Consists of the volunteer standing on one leg while simultaneously stretching the other lower limb in 3 different directions. These are: anterior, posteromedial and posterolateral.
Med Ball Throw | The test will be conducted 3 times: pre-intervention, immediately after the intervention and immediately after training session.
  It involves the volunteer sitting on the floor with their legs apart and having to throw a 2 kg ball forward in front of them.
Close Kinetic Chain Upper Extremity Stability Test | The test will be administered 3 times: pre-intervention, immediately after the intervention and immediately after training session.
  The volunteer assumes a push-up position with their hands 36 inches apart, and their performance is assessed based on how many times in 15 seconds the person can lift one arm

CONTACTS AND LOCATIONS:
Overall Officials: Studnicki, Principal Investigator — Medical University of Gdansk
Locations (1):
- AZS Central Academic Sports Center in Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No